CLINICAL TRIAL: NCT02737592
Title: A Clinical Study to Evaluate the Safety of a Personal Lubricant in Healthy Female Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: ST-7610
Record Dates: First submitted 2016-03-22; First posted 2016-04-14 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Erythema; Edema
MeSH Terms: conditions — Erythema; Edema

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (1):
- Healthy subject (Experimental): Healthy subject exposed to Trojan "Simply Pleasures" Personal Lubricant at least four times weekly for two weeks
  Interventions: Device: Trojan "Simply Pleasure" Personal Lubricant

INTERVENTIONS:
Device: Trojan "Simply Pleasure" Personal Lubricant — silicone base without sensate

SUMMARY:
To evaluate the safety of a personal lubricant when used at least four times weekly for two weeks (including at least twice weekly during sexual intercourse for subjects with monogamous male partners), in a population consisting of healthy females.

ELIGIBILITY:
Inclusion Criteria:

* no participation in a similar study 2-weeks prior
* may be post-menopausal or have had a hysterectomy
* if sexually active, and of child bearing potential, subjects is using adequate non-barrier method of birth control
* free from any vaginal disorders
* sexually active and in a monogamous, heterosexual relationship, and whose male partner is willing and able to give informed consent and agrees to engage in sexual intercourse at least twice each week during the two-week study or is not sexually active
* personal lubricant user and agrees to replace her usual personal lubricant with the investigational product
* can start regardless of where they are in their cycles
* agrees to use the provided investigational product at least four time weekly over the two week study period
* exhibits no clinically significant evidence of vulvar or vaginal irritation, as determined by a study doctor, and no reports of sensory irritation at the baseline exam
* willing to refrain from introducing any new vaginal products, or using vaginal medications or local contraceptives during study
* agrees to refrain from douching or using any medications, powder, lotions or personal care products in the vulvar or perianal area
* willing to use a urine pregnancy test provided to them at baseline and on third visit
* standard medical history form on file
* signed informed consent
* completed HIPAA
* dependable and able to follow directions as outlined
* receives a score of 0 or 0.5 for erythema and edema; and 0 for sensorial irritation (burning, stinging, itching and dryness) during the first examination.

Exclusion Criteria:

* pregnant, nursing or planning a pregnancy
* currently using or has used within two weeks prior to the study initiation, any systemic or topical corticosteroids, vasoconstrictors, antibiotics, anti-inflammatories or antihistamines
* known allergies to vaginal or any cosmetic products
* reports history of recurrent bladder, vaginal infections or incontinence
* exhibits or reports gynecologic abnormalities or has had vaginitis within 60 days prior to study initiation
* uses a vaginal ring, diaphram or cervical/vault caps, condoms, or condoms with spermicide as a means of contraception
* participated in a study involving the vaginal area or in an investigational systemic drug study within two weeks of study initiation
* receives a score higher than 0/5 for erythema, edema or >0 for burning, stinging, or itching, during first examination or shows any other sign of mucosal irregularities

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Laboratories, LLC, Piscataway, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Subject
Started | 34
Completed | 33
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Subject
Number analyzed (Participants) | 33
Age, Customized [Count of Participants; unit: Participants]
  Age 20 - 60 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Observed Local Erythema Based on 5 Point Scale
Description: Number of subjects with observed local erythema by OB/GYN examination as graded on 5 point clinical scale: 0 = normal appearance no irritation, 0.5 = slight, irregular erythema, 1 = mild erythema, 2 = moderate erythema 3 = severe erythema
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Subject
Number analyzed (Participants) | 33
Participants | 0

2. Primary Outcome: Number of Subjects With Observed Edema Based on the 5 Point Scoring Scale
Description: Number of subjects with observed local edema by OB/GYN examination as graded on 5 point clinical scale: 0 = normal appearance no edema, 0.5 = slight edema, 1 = mild edema, 2 = moderate edema 3 = severe edema
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Subject
Number analyzed (Participants) | 33
Participants | 0

ADVERSE EVENTS:
Arm/Group | Healthy Subject
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Master service agreement and confidentiality agreement in place